CLINICAL TRIAL: NCT01983280
Title: The Effect of Healing Touch on Sleep Patterns of Pediatric Burn Patients: A Prospective Cross Over Trial
Brief Title: The Effect of Healing Touch on Sleep Patterns of Pediatric Burn Patients
Acronym: Sleep5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Lois Claire Cone, R.T. (R) (ARRT), HTCP, M. AmSAT, Manager, Radiology, Shriners Hospitals for Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013 6058 09081008
Record Dates: First submitted 2013-09-30; First posted 2013-11-13 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Burn
Keywords: polysomnography; sleep; healing touch; pediatric burn
MeSH Terms: conditions — Burns | interventions — Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healing Touch (Experimental)
  Interventions: Other: Healing Touch

INTERVENTIONS:
Other: Healing Touch

SUMMARY:
Adequate sleep is an important aspect of any healing process, and because it is known that children recovering from burns suffer long term sleep disruptions, the investigators believe that Healing Touch may improve the quality and quantity of sleep in the pediatric burn population.

DETAILED DESCRIPTION:
This study examines the impact of Healing Touch on the quality and quantity of sleep in pediatric burn survivors. Polysomnography recordings are obtained in order to assess nocturnal sleep in conjunction with Healing Touch; which is done on 1 of 2 nights during Polysomnography. Soft background music is played on both nights.

Healing Touch is performed by one of 2 Healing Touch Certified Practitioners.

ELIGIBILITY:
Inclusion Criteria:

1. All pediatric patients (from 5 to 21 years of age) admitted for treatment (following an acute burn injury) to Shriners Hospitals for Children - Cincinnati Burns Hospital will be screened.
2. Include electrical, flame, scald and chemical burns.
3. Signed informed consent

Exclusion Criteria:

1. Patients admitted for treatment unrelated to a burn injury.
2. Patients admitted for less than 2 nights.
3. Patients with face and head grafting if they interfere with the lead placements
4. Neurological disorder

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2009-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Quality of sleep | It takes 1 month for the PSG results to be completed
  Comparison of sleep with and without Healing Touch at bedtime. Polysomnography measures whether the patient enters into all the different stages of sleep, particularly Rapid Eye Movement sleep.

SECONDARY OUTCOMES:
Quantity of sleep | It takes 1 month for the polysomnography results to be completed.
  Polysomnography measures percentages of sleep stages and the overall duration of the combined stages.

CONTACTS AND LOCATIONS:
Locations (1):
- Shriners Hospitals for Children, Cincinnati, Ohio, United States